CLINICAL TRIAL: NCT00905684
Title: Effects of Counseling on the Continuation Rates and Compliance for Newly Prescribed Oral Contraceptives (Yasmin® or Any Other Oral Contraceptives (OC))
Brief Title: Effects of Counseling on the Continuation Rates and Compliance for Newly Prescribed Oral Contraceptives (Yasmin® or Any Other Oral Contraceptives (OC)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer HealthCare AG
Other Study IDs: 14565; YA0801 (Other: Company internal)
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Contraception
Keywords: Compliance; Hormonal Contraception
MeSH Terms: conditions — Patient Compliance | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: EE30/DRSP (Yasmin, BAY86-5131)
- Group 2
  Interventions: Drug: Any other OC

INTERVENTIONS:
Drug: EE30/DRSP (Yasmin, BAY86-5131) — Patients under regular daily life treatment receiving Yasmin according to local drug information
  Groups: Group 1
Drug: Any other OC — Patients under regular daily life treatment receiving any other OC according to local drug information
  Groups: Group 2

SUMMARY:
This study is a prospective, company-sponsored, non-interventional cohort study of up to 5000 patients in European countries and countries in Middle East who are newly prescribed any available OC. Patients will be followed up approximately 6 months after initial visit. Selection of Study Population: Women can be enrolled after decision for treatment with Yasmin or any other OC has been made. Physicians should consult the full prescribing information for the respective OC before enrolling patients and familiarize themselves with the safety information in the product package label.

ELIGIBILITY:
Inclusion Criteria:

* Women who have been found eligible for OC use and have newly been prescribed an OC in accordance with the terms of the respective marketing authorization
* Starter (first-ever user of an OC) and switcher from another OC (incl. women with a history of OC use)

Exclusion Criteria:

* The contraindications and warnings of the Summary of Product Characteristics must be followed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who have been found eligible for OC use and have newly been prescribed an OC in accordance with the terms of the respective marketing authorization Starter (first-ever user of an OC) and switcher from another OC (incl. women with a history of OC use)
Sampling Method: Non-Probability Sample
Enrollment: 5446 (Actual)
Dates: Start 2009-06; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Analyses of continuation rates and compliance stratified by the subject's knowledge on the respective topics and time spent for counseling. | After 3 months and at end of study after approx. 6 months.

SECONDARY OUTCOMES:
Analyses stratified by baseline factors such as age group, presence or absence of cycle disorders, and history of oral contraceptive method will be performed as well. | After 3 months and after approx. 6 months.
Special attention will be paid to serious adverse events and unexpected or unlisted ADRs. | Over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Many Locations, Albania
- Many Locations, Bahrain
- Many Locations, Egypt
- Many Locations, Hungary
- Many Locations, Jordan
- Many Locations, Kenya
- Many Locations, Kuwait
- Many Locations, Lebanon
- Many Locations, North Macedonia
- Many Locations, Oman
- Many Locations, Qatar
- Many Locations, Saudi Arabia
- Many Locations, United Arab Emirates